CLINICAL TRIAL: NCT04990791
Title: Characterisation of a Novel Regimen of Very Low-dose Aspirin Combined With Rivaroxaban in Patients With Chronic Coronary Syndromes: WILL lOWer Dose Aspirin be Better With Rivaroxaban in Patients With Chronic Coronary Syndromes?
Brief Title: WILL lOWer Dose Aspirin be Better With Rivaroxaban in Patients With Chronic Coronary Syndromes?
Acronym: WILLOW CCS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: STH20412
Record Dates: First submitted 2021-06-28; First posted 2021-08-04 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Coronary Syndrome
MeSH Terms: conditions — Angina, Unstable | interventions — Aspirin; Rivaroxaban

STUDY DESIGN:
Intervention Model Description: Randomised controlled open-label crossover study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aspirin 20mg (Other): Aspirin 75 mg OD for 14(-2) days then aspirin 20 mg BD plus rivaroxaban 2.5 mg BD for 14(-2) days then aspirin 75 mg OD plus rivaroxaban 2.5 mg BD
  Interventions: Drug: Aspirin 75mg; Drug: Aspirin 20mg; Drug: Rivaroxaban 2.5 mg
- Asprin 75mg (Other): Aspirin 75 mg OD for 14(-2) days then aspirin 75 mg OD plus rivaroxaban 2.5 mg BD for 14(-2) days then aspirin 20 mg BD plus rivaroxaban 2.5 mg BD
  Interventions: Drug: Aspirin 75mg; Drug: Aspirin 20mg; Drug: Rivaroxaban 2.5 mg

INTERVENTIONS:
Drug: Aspirin 75mg — Aspirin 75mg OD for 14 days
Drug: Aspirin 20mg — Aspirin 20mg BD for 14 days
Drug: Rivaroxaban 2.5 mg — Rivaroxaban 2.5mg BD

SUMMARY:
The trial is a pharmacodynamic study to determine the effect of a novel regimen of aspirin 20 mg BD plus rivaroxaban 2.5 mg BD on haemostasis, fibrin clot dynamics, inflammatory markers, platelet function and arachidonic acid metabolites when compared to standard regimens of aspirin 75 mg OD and aspirin 75 mg OD plus rivaroxaban 2.5 mg BD.

In a randomised open-label three-period crossover design, patient participants receiving aspirin 75 mg OD for secondary prevention of IHD will be randomised 1:1 to receive one of two sequences of aspirin: aspirin 75 mg OD, then aspirin 20 mg BD plus rivaroxaban 2.5 mg BD, then aspirin 75 mg OD plus rivaroxaban 2.5 mg BD; or aspirin 75 mg OD, then aspirin 75 mg OD plus rivaroxaban 2.5 mg BD, then aspirin 20 mg BD plus rivaroxaban 2.5 mg BD.

At the end of each 14(-2) day medication period, they will attend a study visit at which blood and urine samples will be obtained, and bleeding time measured, before and 2 hours after the last dose of IMP of the treatment period. The samples will be tested for fibrin clot dynamics; inflammatory markers and cytokines; prostanoids; and platelet function.

Participants will be transitioned back to standard-of-care aspirin 75 mg OD at the end of the third treatment period and followed up by telephone call 14(-2) days later.

DETAILED DESCRIPTION:
Recruitment Potential participants will be identified through review of the records of the South Yorkshire Cardiothoracic Centre and/or by referral by their clinical team.

Specifically, participants may be approached in the following ways:

1. An invitation letter sent by post in combination with a copy of the participant information sheet. There will be a reply slip which they can return by post, and there will be contact details (telephone and email) for the research team to allow them to respond by these methods too.
2. Directly by telephone. In this case, should they be happy to learn more, they will be sent a copy of the invitation letter, participant information sheet and reply slip by post or email, depending on their preference. If they agree to attend for study screening, they will communicate this to the research team by returning the reply slip by post or email, or by contacting the research team directly using the contact details provided to them.
3. Directly in clinics within the Cardiology and Cardiothoracic Surgery Directorate at Sheffield Teaching Hospitals NHS Foundation Trust, upon referral from their clinical team. In this case they will be provided with a copy of the participant information sheet and, if unable to decide whether they wish to attend for screening or not during the clinic visit, will be signposted to the contact details of the research team to provide their response.

   Potential participants who are interested in taking part in the study will then be contacted by the research team to book a screening appointment.

   Screening

   Screening will occur at visit 1. The following study procedures will be performed, after obtaining written consent for the study:
   * Medical history
   * Physical examination
   * Collection of demographic data
   * Vital signs (pulse, blood pressure and temperature).
   * Height, weight and BMI
   * Recording of any concomitant medication
   * Safety blood tests (13.5 ml blood sample for haematology, clinical chemistry and coagulation)
   * Urinalysis (dipstick), plus urinary pregnancy test if female and of childbearing potential. This will also be checked immediately prior to first rivaroxaban exposure at visit 3.
   * Baseline electrocardiogram

   Consent Written, informed consent, using the current version of the approved designated form for this study, will be obtained prior to any study procedures being carried out. This will be explained and obtained by a medically-qualified member of the research team, listed on the delegation log. Participants will have the chance to read the ICF/PIS for as long as they need, and will be able to ask any questions, prior to signing. Minors and those judged to be without the mental capacity to provide informed consent will not be enrolled into the study.

   Participants will remain free to withdraw at any time from the trial, without giving reasons and without prejudicing his/her further treatment, and will be provided with a contact point where he/she may obtain further information about the trial. Samples collected up to the point of withdrawal will only be used after withdrawal if the participant consents for this, otherwise they will be destroyed. However, data collected up to that point will be used for analysis, and this will be explicitly stated in the participant information sheet and consent form.

   The randomisation scheme

   Participants will be randomised to one of the following two treatment sequences, in a 1:1 fashion:

   (A) Aspirin 75 mg OD for 14(-2) days then aspirin 20 mg BD plus rivaroxaban 2.5 mg BD for 14(-2) days then aspirin 75 mg OD plus rivaroxaban 2.5 mg BD or (B) Aspirin 75 mg OD for 14(-2) days then aspirin 75 mg OD plus rivaroxaban 2.5 mg BD for 14(-2) days then aspirin 20 mg BD plus rivaroxaban 2.5 mg BD

   Baseline data At visit 1
   * Medical history
   * Physical examination
   * Demographic data
   * Vital signs (pulse, blood pressure and temperature)
   * Weight and BMI
   * Concomitant medication
   * Lab safety parameters (full blood count, urea & electrolytes, liver function tests, clotting screen, dipstick urinalysis, urinary pregnancy test if female and of childbearing potential)
   * Electrocardiogram findings At visit 2
   * Vital signs: pulse, blood pressure and temperature
   * Physical examination

   Visit 1 - Screening (Day -21 to 0)

   Screening of subjects and all study-related procedures will take place in the Sheffield Clinical Research Facility, a specialist environment for the conduct of clinical research. The following assessments and procedures will be performed:

   - Full informed consent, including completion of the informed consent form
   * Inclusion/exclusion criteria (see section 6)
   * Medical history
   * Physical examination
   * Demographic data
   * Vital signs: pulse, blood pressure and temperature
   * Weight and BMI
   * Concomitant medication
   * Lab safety (13.5 ml blood sample for haematology; clinical chemistry & coagulation; urinalysis)
   * Electrocardiogram

   Visit 2 (Day 0) - Randomisation
   * Vital signs
   * Physical examination
   * Reconfirm eligibility criteria met (by a medically qualified member of the study team, see section 6) and no withdrawal criteria met (section 7.10)
   * Randomisation
   * Provided with supply of aspirin (aspirin lysine) for periods 1, 2 and 3 (2 boxes of 30 sachets)
   * Dose-preparation training for aspirin (aspirin lysine) 75 mg OD, including supply of written illustrated instructions
   * Issue with participant information card detailing treatment allocation, restrictions during the study and contact details for the research team

   Period 1: 14 (-2) days - Participants will receive aspirin (aspirin lysine) 75 mg OD, but should withhold their dose on the morning of visit 3 (during which the dose will be taken).

   Visit 3 - Period 1: Day 14 (-2)
   * Vital signs
   * Physical examination
   * Adverse event recording
   * Concomitant medication recorded
   * Venous blood sample pre- and 2 hours post-dose for fibrin clot dynamics, inflammatory markers, prostanoids and platelet function
   * Bleeding time pre- and 2 hours post dose
   * Urine sample pre- and 2 hours post-dose for prostanoids
   * IMP compliance check for period 1
   * Dispensing of rivaroxaban 2.5 mg tablets for periods 2 and 3 (total 56 tablets)
   * Urine pregnancy test for women of childbearing potential (must not continue to period 2 if positive)
   * Dose-preparation training for aspirin (aspirin lysine) 20 mg BD if allocated to sequence A, including provision of written instructions

   Period 2: 14(-2) days

   Participants will receive their allocated regimen for period 2 for 14(-2) days:
   * If randomised to sequence A they will receive aspirin (aspirin lysine) 20 mg BD plus rivaroxaban 2.5 mg BD in period 2.
   * If randomised to sequence B they will receive aspirin (aspirin lysine) 75 mg BD plus rivaroxaban 2.5 mg BD in period 2.

   Participants should withhold their dose on the morning of visit 4 (during which the dose will be taken).

   Visit 4 : 14(-2) days into period 2 - Physical examination
   * Adverse event recording
   * Concomitant medication recorded
   * Venous blood sample pre- and 2 hours post-dose for fibrin clot dynamics, inflammatory markers, prostanoids and platelet function
   * Bleeding time pre- and 2 hours post dose
   * Urine sample pre- and 2 hours post-dose for prostanoids
   * IMP compliance recorded for period 2
   * Dose-preparation training for aspirin (aspirin lysine) 75 mg OD if allocated to sequence A or 20 mg BD if sequence B, including provision of written instructions

   Period 3: 14(-2) days

   Participants will receive their allocated regimen for period 3 for 14(-2) days:
   * If randomised to sequence A they will receive aspirin (aspirin lysine) 75 mg OD plus rivaroxaban 2.5 mg BD in period 3.
   * If randomised to sequence B they will receive aspirin (aspirin lysine) 20 mg BD plus rivaroxaban 2.5 mg BD in period 3.

   Visit 5 : 14(-2) days into period 3 - Vital signs

   - Physical examination

   - Adverse event recording

   - Concomitant medication recorded

   - Venous blood sample pre- and 2 hours post-dose for fibrin clot dynamics, inflammatory markers, prostanoids and platelet function

   - Bleeding time pre- and 2 hours post dose

   - Urine sample pre- and 2 hours post-dose for prostanoids

   - IMP compliance recorded for period 3
   * Collect and return unused medication to pharmacy
   * Transition to standard of care aspirin 75 mg OD, ensuring participant has a supply of this

   Visit 6 : 14(-2) days after visit 5 (Telephone call) - Telephone follow-up for adverse events and concomitant medication

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures
2. Male or female aged greater than 18 years
3. Existing diagnosis of a chronic coronary syndrome:

   (i) History of stable angina or (ii) History of an acute coronary syndrome event >1 year ago or (iii) Previous evidence on imaging of either at least one stenosis >50% in an epicardial coronary artery or a myocardial perfusion defect
4. Receiving single antiplatelet therapy with aspirin 75 mg once daily

Exclusion Criteria:

1. Any history of haemorrhagic stroke or lacunar stroke
2. History of ischaemic stroke or transient ischaemic attack in the last year
3. Heart failure associated with NYHA class III or IV symptoms
4. Estimated glomerular filtration rate <15 ml/min
5. Planned procedure for coronary revascularization
6. Any planned surgery or other procedure that may require suspension or discontinuation of antiplatelet therapy expected to occur within 3 months of randomisation
7. Prior intention by patient or physician to discontinue aspirin within the study period
8. Receiving doses of aspirin other than 75 mg once daily
9. Treatment or planned treatment with antiplatelet medication apart from aspirin (eg. clopidogrel, prasugrel, ticagrelor, dipyridamole, ticlopidine)
10. Current use of a loop, thiazide or potassium sparing diuretic (affects prostanoid assays)
11. Any acute coronary syndrome event, percutaneous coronary intervention or coronary artery bypass grafting within 1 year prior to randomisation
12. Current or planned use of an oral anticoagulant (e.g. warfarin, dabigatran, rivaroxaban [including 2.5 mg BD], apixaban, edoxaban) or parenteral anticoagulant (eg. unfractionated heparin, low molecular weight heparin, bivalirudin)
13. Current or planned use of a GPIIb/IIIa inhibitor (eg. abciximab, tirofiban)
14. Current or planned use of a fibrinolytic agent (eg. tissue plasminogen activator)
15. Requiring or likely to require treatment with a non-steroidal anti-inflammatory drug (NSAID), including COX2 inhibitors, and including regular or intermittent/as required use
16. Current or planned use of a strong CYP3A4 inhibitor (eg, ketoconazole, itraconazole, voriconazole, telithromycin, clarithromycin [but not erythromycin or azithromycin], nefazadone, ritonavir, saquinavir, nelfinavir, indinavir, atanazavir, cobicistat or over 1 litre daily of grapefruit juice), strong inducer (e.g. rifampin/rifampicin, rifabutin, phenytoin, carbamazepine, phenobarbital), a selective serotonin reuptake inhibitor (SSRI) or selective noradrenergic reuptake inhibitor (SNRI).
17. Clinically significant liver disease, defined as known or suspected diagnosis of hepatic cirrhosis with current Child Pugh class B or C; or elevation of serum alanine transferase or aspartate transferase greater than 3 times the upper limit of the normal range for the processing laboratory.
18. History of alcohol or drug abuse, defined as regular use of an illicit substance for recreational purposes or regular consumption of greater than 50 units (males) or 35 units (females) of alcohol per week, in the last year
19. Co-morbidity associated with life expectancy less than 1 year
20. Any other condition deemed by the investigator to significantly affect haemostasis, coagulation, bleeding risk or ability to comply with the study protocol.
21. Females of child-bearing potential unless negative pregnancy test at screening and willing to use effective contraception (i.e. established use of oral, injected or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS) or barrier methods of contraception with spermicide or sole male partner with prior vasectomy and confirmed absence of sperm in ejaculate) for the duration of treatment with study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-08-26 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Bleeding Time Difference | Until 14 (-2) days after last IMP dose
  The primary endpoint will be difference in bleeding time, measured at 2 hours post-dose, assessed between aspirin (aspirin lysine) 75 mg once-daily alone vs. aspirin (aspirin lysine) 20 mg twice-daily plus rivaroxaban 2.5 mg twice-daily and aspirin (aspirin lysine) 75 mg once-daily alone vs. aspirin (aspirin lysine) 75 mg once-daily plus rivaroxaban 2.5 mg twice-daily.

SECONDARY OUTCOMES:
Bleeding time pre-dose | Until 14 (-2) days after last IMP dose
  A secondary endpoint will be the difference in bleeding time measured at pre-dose
Fibrin clot lag time by fibrin clot turbidimetry | Until 14 (-2) days after last IMP dose
  A secondary endpoint will be the difference in fibrin clot lag time at pre-dose and 2 hours post-dose
Fibrin clot lysis time by fibrin clot turbidimetry | Until 14 (-2) days after last IMP dose
  A secondary endpoint will be the difference in fibrin lysis lag time at pre-dose and 2 hours post-dose
Plasma TNF by enzyme-linked immunosorbent assay (ELISA)/multiplex bead assay (MBA) | Until 14 (-2) days after last IMP dose
  A secondary endpoint will be the difference in Plasma TNF-α at pre-dose and 2 hours post-dose
Plasma IL-6 by ELISA | Until 14 (-2) days after last IMP dose
  A secondary endpoint will be the difference in Plasma IL-6 at pre-dose and 2 hours post-dose
Serum CRP (Roche Cobas assay) | Until 14 (-2) days after last IMP dose
  A secondary endpoint will be the difference in Serum CRP at 2 hours post-dose
Leukocyte count (and subsets), by automated cell counting | Until 14 (-2) days after last IMP dose
  A secondary endpoint will be the difference in Leukocyte count at pre-dose and 2 hours post-dose
Serum TXB2 by ELISA | Until 14 (-2) days after last IMP dose
  A secondary endpoint will be the difference in Serum TXB2 at pre-dose and 2 hours post-dose
Urine PGI-M by ELISA | Until 14 (-2) days after last IMP dose
  A secondary endpoint will be the difference in Urine PGI-M at pre-dose and 2 hours post-dose
Urine TxM by ELISA | Until 14 (-2) days after last IMP dose
  A secondary endpoint will be the difference in Urine TxM at pre-dose and 2 hours post-dose
Platelet aggregation responses to AA, collagen and adenosine diphosphate ADP by light transmittance aggregometry | Until 14 (-2) days after last IMP dose
  Mean platelet aggregation responses to arachidonic acid (AA), collagen and adenosine diphosphate (ADP), at pre-dose and 2 hours post-dose
Final clot turbidity by fibrin clot turbidimetry | Until 14 (-2) days after last IMP dose
  A secondary endpoint will be the final clot turbidity at pre-dose and 2 hours post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The data arising from the trial will be owned by University of Sheffield and will not be disseminated to other researchers

REFERENCES:
- [Background] Task Force Members; Montalescot G, Sechtem U, Achenbach S, Andreotti F, Arden C, Budaj A, Bugiardini R, Crea F, Cuisset T, Di Mario C, Ferreira JR, Gersh BJ, Gitt AK, Hulot JS, Marx N, Opie LH, Pfisterer M, Prescott E, Ruschitzka F, Sabate M, Senior R, Taggart DP, van der Wall EE, Vrints CJ; ESC Committee for Practice Guidelines; Zamorano JL, Achenbach S, Baumgartner H, Bax JJ, Bueno H, Dean V, Deaton C, Erol C, Fagard R, Ferrari R, Hasdai D, Hoes AW, Kirchhof P, Knuuti J, Kolh P, Lancellotti P, Linhart A, Nihoyannopoulos P, Piepoli MF, Ponikowski P, Sirnes PA, Tamargo JL, Tendera M, Torbicki A, Wijns W, Windecker S; Document Reviewers; Knuuti J, Valgimigli M, Bueno H, Claeys MJ, Donner-Banzhoff N, Erol C, Frank H, Funck-Brentano C, Gaemperli O, Gonzalez-Juanatey JR, Hamilos M, Hasdai D, Husted S, James SK, Kervinen K, Kolh P, Kristensen SD, Lancellotti P, Maggioni AP, Piepoli MF, Pries AR, Romeo F, Ryden L, Simoons ML, Sirnes PA, Steg PG, Timmis A, Wijns W, Windecker S, Yildirir A, Zamorano JL. 2013 ESC guidelines on the management of stable coronary artery disease: the Task Force on the management of stable coronary artery disease of the European Society of Cardiology. Eur Heart J. 2013 Oct;34(38):2949-3003. doi: 10.1093/eurheartj/eht296. Epub 2013 Aug 30. No abstract available. PMID 23996286
- [Background] Knuuti J, Wijns W, Saraste A, Capodanno D, Barbato E, Funck-Brentano C, Prescott E, Storey RF, Deaton C, Cuisset T, Agewall S, Dickstein K, Edvardsen T, Escaned J, Gersh BJ, Svitil P, Gilard M, Hasdai D, Hatala R, Mahfoud F, Masip J, Muneretto C, Valgimigli M, Achenbach S, Bax JJ; ESC Scientific Document Group. 2019 ESC Guidelines for the diagnosis and management of chronic coronary syndromes. Eur Heart J. 2020 Jan 14;41(3):407-477. doi: 10.1093/eurheartj/ehz425. No abstract available. PMID 31504439
- [Background] Eikelboom JW, Connolly SJ, Bosch J, Dagenais GR, Hart RG, Shestakovska O, Diaz R, Alings M, Lonn EM, Anand SS, Widimsky P, Hori M, Avezum A, Piegas LS, Branch KRH, Probstfield J, Bhatt DL, Zhu J, Liang Y, Maggioni AP, Lopez-Jaramillo P, O'Donnell M, Kakkar AK, Fox KAA, Parkhomenko AN, Ertl G, Stork S, Keltai M, Ryden L, Pogosova N, Dans AL, Lanas F, Commerford PJ, Torp-Pedersen C, Guzik TJ, Verhamme PB, Vinereanu D, Kim JH, Tonkin AM, Lewis BS, Felix C, Yusoff K, Steg PG, Metsarinne KP, Cook Bruns N, Misselwitz F, Chen E, Leong D, Yusuf S; COMPASS Investigators. Rivaroxaban with or without Aspirin in Stable Cardiovascular Disease. N Engl J Med. 2017 Oct 5;377(14):1319-1330. doi: 10.1056/NEJMoa1709118. Epub 2017 Aug 27. PMID 28844192
- [Background] Sumaya W, Wallentin L, James SK, Siegbahn A, Gabrysch K, Bertilsson M, Himmelmann A, Ajjan RA, Storey RF. Fibrin clot properties independently predict adverse clinical outcome following acute coronary syndrome: a PLATO substudy. Eur Heart J. 2018 Apr 1;39(13):1078-1085. doi: 10.1093/eurheartj/ehy013. PMID 29390064
- [Background] Konigsbrugge O, Weigel G, Quehenberger P, Pabinger I, Ay C. Plasma clot formation and clot lysis to compare effects of different anticoagulation treatments on hemostasis in patients with atrial fibrillation. Clin Exp Med. 2018 Aug;18(3):325-336. doi: 10.1007/s10238-018-0490-9. Epub 2018 Feb 7. PMID 29417256
- [Background] Patrono C, Morais J, Baigent C, Collet JP, Fitzgerald D, Halvorsen S, Rocca B, Siegbahn A, Storey RF, Vilahur G. Antiplatelet Agents for the Treatment and Prevention of Coronary Atherothrombosis. J Am Coll Cardiol. 2017 Oct 3;70(14):1760-1776. doi: 10.1016/j.jacc.2017.08.037. PMID 28958334
- [Background] Patrono C. Aspirin as an antiplatelet drug. N Engl J Med. 1994 May 5;330(18):1287-94. doi: 10.1056/NEJM199405053301808. No abstract available. PMID 8145785
- [Background] Ajjan RA, Standeven KF, Khanbhai M, Phoenix F, Gersh KC, Weisel JW, Kearney MT, Ariens RA, Grant PJ. Effects of aspirin on clot structure and fibrinolysis using a novel in vitro cellular system. Arterioscler Thromb Vasc Biol. 2009 May;29(5):712-7. doi: 10.1161/ATVBAHA.109.183707. Epub 2009 Mar 12. PMID 19286636
- [Background] Kiers D, van der Heijden WA, van Ede L, Gerretsen J, de Mast Q, van der Ven AJ, El Messaoudi S, Rongen GA, Gomes M, Kox M, Pickkers P, Riksen NP. A randomised trial on the effect of anti-platelet therapy on the systemic inflammatory response in human endotoxaemia. Thromb Haemost. 2017 Aug 30;117(9):1798-1807. doi: 10.1160/TH16-10-0799. Epub 2017 Jul 6. PMID 28692111
- [Background] Thomas MR, Outteridge SN, Ajjan RA, Phoenix F, Sangha GK, Faulkner RE, Ecob R, Judge HM, Khan H, West LE, Dockrell DH, Sabroe I, Storey RF. Platelet P2Y12 Inhibitors Reduce Systemic Inflammation and Its Prothrombotic Effects in an Experimental Human Model. Arterioscler Thromb Vasc Biol. 2015 Dec;35(12):2562-70. doi: 10.1161/ATVBAHA.115.306528. Epub 2015 Oct 29. PMID 26515417
- [Background] Ridker PM, Everett BM, Thuren T, MacFadyen JG, Chang WH, Ballantyne C, Fonseca F, Nicolau J, Koenig W, Anker SD, Kastelein JJP, Cornel JH, Pais P, Pella D, Genest J, Cifkova R, Lorenzatti A, Forster T, Kobalava Z, Vida-Simiti L, Flather M, Shimokawa H, Ogawa H, Dellborg M, Rossi PRF, Troquay RPT, Libby P, Glynn RJ; CANTOS Trial Group. Antiinflammatory Therapy with Canakinumab for Atherosclerotic Disease. N Engl J Med. 2017 Sep 21;377(12):1119-1131. doi: 10.1056/NEJMoa1707914. Epub 2017 Aug 27. PMID 28845751
- [Background] Teng R, Maya J, Butler K. Evaluation of the pharmacokinetics and pharmacodynamics of ticagrelor co-administered with aspirin in healthy volunteers. Platelets. 2013;24(8):615-24. doi: 10.3109/09537104.2012.748185. Epub 2012 Dec 18. PMID 23249161
- [Background] Choi J, Hwang SY, Ahn K. Interplay between RNASEH2 and MOV10 controls LINE-1 retrotransposition. Nucleic Acids Res. 2018 Feb 28;46(4):1912-1926. doi: 10.1093/nar/gkx1312. PMID 29315404
- [Background] Ghys T, Malfait R, VAN den Bossche J. Performance evaluation of the Sysmex XS-1000i automated haematology analyser. Int J Lab Hematol. 2009 Oct;31(5):560-6. doi: 10.1111/j.1751-553X.2008.01081.x. Epub 2009 Jun 18. PMID 18616754
- [Background] Parker WAE, Orme RC, Hanson J, Stokes HM, Bridge CM, Shaw PA, Sumaya W, Thorneycroft K, Petrucci G, Porro B, Judge HM, Ajjan RA, Rocca B, Storey RF. Very-low-dose twice-daily aspirin maintains platelet inhibition and improves haemostasis during dual-antiplatelet therapy for acute coronary syndrome. Platelets. 2019;30(2):148-157. doi: 10.1080/09537104.2019.1572880. Epub 2019 Feb 13. PMID 30759035
- [Background] Doroszko A, Szahidewicz-Krupska E, Janus A, Jakubowski M, Turek A, Ilnicka P, Szuba A, Mazur G, Derkacz A. Endothelial dysfunction in young healthy men is associated with aspirin resistance. Vascul Pharmacol. 2015 Apr-Jun;67-69:30-7. doi: 10.1016/j.vph.2015.02.001. Epub 2015 Feb 17. PMID 25697550
- [Background] Olson MT, Kickler TS, Lawson JA, McLean RC, Jani J, FitzGerald GA, Rade JJ. Effect of assay specificity on the association of urine 11-dehydro thromboxane B2 determination with cardiovascular risk. J Thromb Haemost. 2012 Dec;10(12):2462-9. doi: 10.1111/jth.12026. PMID 23072449
- [Background] Sanchez A, Mirabel JL, Barrenechea E, Eugui J, Puelles A, Castaneda A. Evaluation of an improved immunoturbidimetic assay for serum C-reactive protein on a COBAS INTEGRA 400 Analyzer. Clin Lab. 2002;48(5-6):313-7. PMID 12071582
- [Background] Harrell FE Jr, Lee KL, Matchar DB, Reichert TA. Regression models for prognostic prediction: advantages, problems, and suggested solutions. Cancer Treat Rep. 1985 Oct;69(10):1071-77. PMID 4042087